CLINICAL TRIAL: NCT00637325
Title: TOP Trial. A Randomised Phase III Clinical Trial of Trastuzumab (Herceptin) Optimization in Patients With Locally Advanced and/or Metastatic Breast Cancer Overexpressing HER2 After a First Line Chemotherapy Plus Trastuzumab.
Brief Title: Trastuzumab Optimization Trial in Breast Cancer
Acronym: TOP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regione Lombardia (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other); Istituto Clinico Humanitas (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOP
Record Dates: First submitted 2008-03-07; First posted 2008-03-17 (Estimated); Last update posted 2008-03-17 (Estimated); Status verified 2008-03

CONDITIONS: Metastatic or Locally Advanced Breast Cancer
Keywords: trastuzumab optimization in breast cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Trastuzumab

ARMS (2):
- A (Experimental): In the maintenance study:
  ARM A: maintenance of trastuzumab
  In the 2nd line study:
  ARM A: trastuzumab plus chemotherapy treatment
  Interventions: Drug: trastuzumab
- B (No Intervention): In the maintenance study:
  ARM B: interruption of trastuzumab treatment
  In the 2nd line study:
  ARM B: chemotherapy alone

INTERVENTIONS:
Drug: trastuzumab — In the maintenance study trastuzumab will be administrated once every 3 weeks at the dose of 6 mg/kg by intravenous infusion over 90 minutes until progression of disease. In the 2nd line study, to accomplish the schedule of concomitant second line chemotherapy, trastuzumab will be given on a weekly (2 mg/kg) or a 3-weekly (6 mg/kg).
  Other Names: Herceptin
  Arms: A

SUMMARY:
This is an open-label, randomised phase III, multicentre, Italian study designed to investigate the role of trastuzumab in patients with locally advanced and/or metastatic breast cancer over expressing HER2 who received a first line chemotherapy containing trastuzumab. The trial in divided in two studies: 1. The maintenance study will be conducted in patients not progressing to a first line chemotherapy plus trastuzumab. 2. The 2nd line study will be conducted in patients progressing to a first line chemotherapy plus trastuzumab.

DETAILED DESCRIPTION:
This project consists of two independent, following specific eligibility criteria and different randomisation schemes studies, later on called maintenance study and 2nd line study. All patients enrolled in the maintenance study, after disease progression should be screened to enter the 2nd line study. Maintenance study: Open-label, randomised, phase III, multicenter, Italian study designed to investigate the role of a maintenance therapy with trastuzumab in patients with locally advanced and/or metastatic breast cancer over expressing HER2 and not progressed to a first line chemotherapy plus trastuzumab. Patients will be ed to: Arm A: maintenance of trastuzumab treatment Arm B: interruption of trastuzumab treatment with a ratio 2 maintenance trastuzumab : 1 interruption of trastuzumab. Trastuzumab will be administered intravenously once every 3 weeks until progression of disease, unmanageable toxicity or patient refusal. Patients will be evaluated for progression every 9 weeks (corresponding to the time required to complete the evaluation after every 3 trastuzumab infusions). For patients whose disease has not progressed two years after enrolment, treatment will continue according to physician decision and disease assessments will be made following the routine clinical practice. Follow-up will be continued until the achievement of the required number of events. 2nd line study: Open-label, randomised, phase III, multicentre, Italian study designed to investigate the role of a second line therapy with trastuzumab in patients with locally advanced and/or metastatic breast cancer over expressing HER2 and progressed to a first line chemotherapy plus trastuzumab. Patients will be randomised to: Arm A: trastuzumab + chemotherapy treatment Arm B: chemotherapy alone with a ratio 1 trastuzumab + chemotherapy treatment : 1 chemotherapy alone. Trastuzumab will be administered intravenously, concomitant to a second line chemotherapy of physician's choice. Trastuzumab can be given on a weekly or 3-weekly schedule to accomplish the schedule of concomitant chemotherapy, until progression of disease, unmanageable toxicity or patient refusal. Patients will be evaluated for progression every 9 weeks (corresponding to the time required to complete the evaluation after every 3 trastuzumab infusions). Follow-up will be continued until the achievement of the required number of events. In maintenance study, trastuzumab will be given in an outpatient setting every 3 weeks at the dose of 6 mg/Kg by intravenous infusion over 90 minutes, or over 30 minutes at the Investigator's discretion followed by 30 minutes observation time. If the last previous dose of trastuzumab was given more than 4 weeks before entering the study, patients will receive a re-loading dose of trastuzumab 8 mg/kg over 90 minutes, followed by 30 minutes observation time. Therapy with trastuzumab will continue until progression of disease, unmanageable toxicity or patient refusal. For patients whose disease has not progressed two years after enrolment, treatment will continue according to physician decision and disease assessments will be made following the routine clinical practice. In 2nd line study, to accomplish the schedule of concomitant second line chemotherapy, trastuzumab will be given on a weekly (2 mg/kg) or a 3-weekly (6 mg/kg) basis with the modalities of the maintenance study, according to clinician's decision. Concomitant second line chemotherapy will be left at physician's choice. If the last previous dose of trastuzumab was given more than 4 weeks before entering the study, patients will receive a re-loading dose of trastuzumab 4 mg/kg over 60 minutes, followed by 30 minutes observation time.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age. Patients older of 70 years of age are eligible on the basis of an individual risk-benefit assessment by the investigator
* Histologically confirmed breast cancer with locally advanced and/or metastatic disease
* Over expression of HER2 (3+) as determined by IHC or amplification of HER2/c-erbB2 by FISH/CISH of the primary tumour or of a metastasis
* Assessable disease. The presence of measurable disease is not needed for enrolment. Patients with bone lesions, ascites and pleural effusion as only sites of disease are considered eligible
* Completion of a first line chemotherapy in association with trastuzumab given for at least 6 months for advanced disease. The last dose of trastuzumab should have to be given within 6 weeks prior to randomisation for treatments given with a 3 weekly schedule or within 3 weeks if a weekly schedule was used (only for maintenance study)
* Progressive disease during or within 6 months from the completion of a first line chemotherapy plus trastuzumab for advanced disease or within 6 months from the completion of an adjuvant treatment for early disease (only for 2nd line study). Patients progressing more than 6 months after the completion of a first line trastuzumab-containing regimen should be re-treated with the previous regimen and included in 2nd line study after evidence of progression.
* Signed written informed consent obtained prior to any study specific study procedures

Exclusion Criteria:

* ECOG-PS >2
* Pregnant or lactating women. Women of childbearing potential must implement adequate contraceptive measures
* Previous or current malignancies at other sites, with the exception of adequately treated in situ carcinoma of the cervix uteri, basal or squamous cell carcinoma of the skin, or other cancer curatively treated by surgery and with no evidence of disease for at least 5 years.
* Baseline LVEF <50% (measured by echocardiography or MUGA) performed within 4 weeks prior to randomisation. History of documented congestive heart failure, angina pectoris requiring antianginal medication, evidence of transmural infarction ECG, poorly controlled hypertension (systolic > 180 mmHg or diastolic > 100 mmHg); clinically significant valvular heart disease; high-risk uncontrolled arrhythmias
* Presence of CNS metastases, not amenable to curative therapy. Patients with previously treated CNS metastases must be asymptomatic and stable at radiological imaging from at least 3 months
* Patients with dyspnoea at rest due to malignant or other disease, or who require supportive oxygen therapy. Patients with pre-existing lung disease or advanced pulmonary involvement may be at increased risk of serious toxicities with trastuzumab and should be evaluated carefully before entry into the study
* Concomitant chemotherapy with anthracyclines, including liposomal drugs (only for 2nd line study)
* Treatment with any investigational drug within 30 days before beginning of enrolment in the trial
* History or presence of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of trastuzumab

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-05 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
progression free survival for maintenance study and overall survival for 2nd line study | 2.5 years

SECONDARY OUTCOMES:
overall survival for the maintenance study and progression free survival for the 2nd line study | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (25):
- Italy (25):
  - Ospedale E. Profili, Fabriano, Ancona
  - Humanitas Cliniche Gavazzeni, Bergamo, Bergamo
  - Azienda Ospedaliera Treviglio- Caravaggio, Treviglio, Bergamo
  - Policlinico Sant'Orsola - Malpighi, Bologna, Bologna
  - Ospedale Sant'Orsola Fatebenefratelli, Brescia, Brescia
  - Ospedale A. Perrino, Brindisi, Brindisi
  - Policlinico Universitario, Monserrato, Cagliari
  - Azienda Ospedaliera Sant' Anna, Como, Como
  - Azienda Ospedaliera Istituti Ospitalieri, Cremona, Cremona
  - Ospedale Alessandro Manzoni, Lecco, Lecco
  - Azienda Ospedaliera di Melegnano - Presidio Ospedaliero di Gorgonzola, Gorgonzola, Milano
  - Ospedale Fatebenefratelli e Oftalmico, Milan, MIlano
  - Fondazione San Raffaele del Monte Tabor, Milan, MIlano
  - Istituto Europeo di Oncologia, Milan, Milano
  - Azienda Ospedaliera San Paolo, Milan, Milano
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Azienda Ospedaliero-Universitaria di Parma, Parma, Parma
  - Azienda Ospedaliera Ospedale San Salvatore, Pesaro, Pesaro - Urbino
  - Ospedale Santa Croce, Fano, Pesaro-Urbino
  - Ospedale Misericordia e Dolce - USL 4, Prato, Prato
  - Dipartimento Oncologico USL 7 Siena, Siena, Siena
  - Ospedale E. Morelli, Sondalo, Sondrio
  - Ospedale Civile di Sondrio, Sondrio, Sondrio
  - Azienda Ospedaliera Busto Arsizio - Presidio ospedaliero Saronno, Saronno, Varese
  - Ospedale "Di Circolo e Fonadazione Macchi", Varese, Varese